CLINICAL TRIAL: NCT01673217
Title: A Phase I Clinical Trial of NY-ESO-1 Protein Immunization in Combination With 5-AZA-2'-Deoxycytidine (Decitabine) in Patients Receiving Liposomal Doxorubicin for Recurrent Epithelial Ovarian or Primary Peritoneal Carcinoma
Brief Title: Decitabine, Vaccine Therapy, and Pegylated Liposomal Doxorubicin Hydrochloride in Treating Patients With Recurrent Ovarian Epithelial Cancer, Fallopian Tube Cancer, or Peritoneal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 127008; NCI-2010-00105 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCT00887796 (obsolete NCT alias)
Record Dates: First submitted 2012-08-22; First posted 2012-08-27 (Estimated); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Recurrent Fallopian Tube Cancer; Recurrent Ovarian Epithelial Cancer; Recurrent Primary Peritoneal Cavity Cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Decitabine; liposomal doxorubicin; sargramostim; Granulocyte-Macrophage Colony-Stimulating Factor; incomplete Freund's adjuvant; montanide ISA 51; Immunohistochemistry; Chromatography, Liquid; Mass Spectrometry; Reverse Transcriptase Polymerase Chain Reaction; DNA Methylation; Enzyme-Linked Immunosorbent Assay

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (chemotherapy and vaccine therapy) (Experimental): Patients receive decitabine IV over 3 hours on day 1, pegylated liposomal doxorubicin hydrochloride IV on day 8, and NY-ESO-1 peptide vaccine emulsified in incomplete Freund's adjuvant and sargramostim subcutaneously on day 15. Treatment repeats every 28 days for 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: decitabine; Biological: NY-ESO-1 peptide vaccine; Drug: pegylated liposomal doxorubicin hydrochloride; Biological: sargramostim; Biological: incomplete Freund's adjuvant; Other: immunohistochemistry staining method; Other: liquid chromatography; Other: mass spectrometry; Genetic: reverse transcriptase-polymerase chain reaction; Other: laboratory biomarker analysis; Genetic: DNA methylation analysis; Other: enzyme-linked immunosorbent assay

INTERVENTIONS:
Drug: decitabine — Given IV
  Other Names: 5-aza-dCyd; 5AZA; DAC
Biological: NY-ESO-1 peptide vaccine — Given SC
  Other Names: ESO-1 Peptide Vaccine
Drug: pegylated liposomal doxorubicin hydrochloride — Given IV
  Other Names: CAELYX; Dox-SL; DOXIL; doxorubicin hydrochloride liposome; LipoDox
Biological: sargramostim — Given SC
  Other Names: GM-CSF; Leukine; Prokine
Biological: incomplete Freund's adjuvant — Given SC
  Other Names: IFA; ISA-51; Montanide ISA 51
Other: immunohistochemistry staining method — Correlative studies
  Other Names: immunohistochemistry
Other: liquid chromatography — Correlative studies
  Other Names: LC
Other: mass spectrometry — Correlative studies
Genetic: reverse transcriptase-polymerase chain reaction — Correlative studies
  Other Names: RT-PCR
Other: laboratory biomarker analysis — Correlative studies
Genetic: DNA methylation analysis — Correlative studies
Other: enzyme-linked immunosorbent assay — Correlative studies
  Other Names: ELISA

SUMMARY:
This phase I trial is studying the side effects and best dose of decitabine when given together with pegylated liposomal doxorubicin hydrochloride and vaccine therapy in treating patients with recurrent ovarian epithelial cancer, fallopian tube cancer, or peritoneal cancer. Drugs used in chemotherapy, such as decitabine and pegylated liposomal doxorubicin hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Vaccines made from a peptide or antigen may help the body build an effective immune response to kill tumor cells. Giving combination chemotherapy together with vaccine therapy may kill more tumor cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety of 5-aza-2'-deoxycytidine (decitabine) in combination with immunization with NYESO-I protein mixed with montanide and granulocyte-macrophage colony stimulating factor (GM-CSF) in patients scheduled to receive liposomal doxorubicin for recurrent epithelial ovarian, fallopian tube or primary peritoneal carcinoma.

SECONDARY OBJECTIVES:

I. To evaluate NY-ESO-l specific cellular and humoral immunity by determination of NY-ESO-I specific antibody, CD8+ and CD4+ T-cells following immunization with NY-ESO-l protein mixed with montanide and GM-CSF in combination with 5-aza-2' -deoxycytidine (decitabine) in patients receiving liposomal doxorubicin for recurrent epithelial ovarian, fallopian tube or primary peritoneal carcinoma.

II. To determine the impact of 5-aza-2'-deoxycytidine on NY-ESO-I specific expression, NY-ESO-l promoter methylation, and global DNA methylation.

III. To compare the time to progression (ttp) for the proposed therapy with the ttp for standard therapy (historical studies).

OUTLINE: This is a dose escalation study of decitabine.

Patients receive decitabine intravenously (IV) over 3 hours on day 1, pegylated liposomal doxorubicin hydrochloride IV on day 8, and NY-ESO-1 peptide vaccine emulsified in incomplete Freund's adjuvant and sargramostim subcutaneously on day 15. Treatment repeats every 28 days for 4 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with relapsed epithelial ovarian cancer (including fallopian tube and primary peritoneal cancer) who will receive liposomal doxorubicin as salvage therapy for recurrent disease
* Patients may have received up to four previous lines of chemotherapy
* The relapse may be defined by an increase in CA125; there may or may not be either measurable or symptomatic disease
* Any human leukocyte antigen (HLA) type
* No requirement for tumor expression of NY-ESO-1
* Karnofsky performance status of > 70%
* Not previously treated with doxorubicin
* Life expectancy >= 6 months
* Hematology and biochemistry laboratory results within the limits normally expected for the patient population, without evidence of major organ failure
* No immunodeficiency
* Have been informed of other treatment options
* Able and willing to give valid written informed consent
* Neutrophil count >= 1.5 x 10^9
* Platelet count >= 100 x 10^9
* Serum creatinine =< 2.1 mg/dL
* Serum bilirubin =< 2 mg/dL
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 2.6 x upper limit of normal (ULN) (normal ranges: AST 15-46 U/L; ALT 11-66 U/L)

Exclusion Criteria:

* Metastatic disease to the central nervous system for which other therapeutic options, including radiotherapy, may be available
* Other serious illnesses (e.g., serious infections requiring antibiotics, bleeding disorders)
* History of autoimmune disease (e.g., thyroiditis, lupus) except vitiligo
* Concomitant systemic treatment with corticosteroids, anti-histamine or non-steroidal anti-inflammatory drugs; specific CQX-2 inhibitors are permitted
* Chemotherapy, radiation therapy, or immunotherapy within 4 weeks prior to first dosing of study agent (6 weeks for nitrosoureas)
* Known human immunodeficiency virus (HIV) positivity
* Known allergy or history of life threatening reaction to GM-CSF
* Myocardial infarction, angina, congestive heart failure, cardiomyopathy, stroke or transient ischemic attack, chest pain or shortness of breath with activity, or other heart conditions being treated by a doctor
* Participation in any other clinical trial involving another investigational agent within 4 weeks prior to first dosing of study agent
* Mental impairment that may compromise the ability to give informed consent and comply with the requirements of the study
* Lack of availability of a patient for immunological and clinical follow-up assessment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2009-04; Primary Completion 2011-10 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Toxicity as assessed by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v3.0 | Up to 6 months
  Estimated with a one-sided, 95%, Wilson score binomial confidence interval.

SECONDARY OUTCOMES:
NY-ESO-1 specific cellular and humoral immunity as assessed by NY-ESO-1-specific CD8+ and CD4+ T cells and antibodies and frequency of CD4+ CD25+ FOXP3+ regulatory T cells | Up to 6 months
  Will be summarized by quartiles. Also, confidence intervals will be constructed for the median and the mean.
NY-ESO-l expression using Q-RT-PCR and IHC | Days 1, 8, 15, 36, 43, 64, 71, 92, and 99
Time to progression | Up to 6 months
  Summarized by a Kaplan-Meier survival curve.
NY-ESO-l promoter DNA methylation using pyrosequencing | Days 1, 8, 15, 36, 43, 64, 71, 92, and 99
Global genomic DNA methylation using liquid chromatography-mass spectrometry (LC-MS) and LINE-l pyrosequencing | Days 1, 8, 15, 36, 43, 64, 71, 92, and 99

CONTACTS AND LOCATIONS:
Overall Officials: Kunle Odunsi, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States